CLINICAL TRIAL: NCT02115308
Title: Characterization of Changes in Ventricular Mechanics in Response to Lexiscan Stress Using Tagged Cine Cardiac Magnetic Resonance Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Timothy M. Bateman (Other)
Collaborators: Saint Luke's Health System (Other); Saint Luke's Cardiovascular Consultants (Other)
Responsible Party: Sponsor-Investigator, Timothy M. Bateman, Medical Director, Aspire Foundation
Organization: Aspire Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Astellas CMR Tagging
Record Dates: First submitted 2014-04-01; First posted 2014-04-16 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regadenoson (Other): Regadenoson is a single-use, pre-filled syringe containing 0.4 mg/5 mL of regadenoson.
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — Regadenoson injection is a pharmacologic stress agent indicated for radionuclide myocardial perfusion imaging.
  Other Names: Lexiscan

SUMMARY:
The purpose of this study is to measure the changes in cardiac function during a Lexiscan pharmacologic stress test using cardiac magnetic resonance imaging test.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial rest/regadenoson stress perfusion PET study within 60 days
* Normal rest LVEF (greater than or equal to 50%)
* No change in symptoms or treatment between the PET and the MRI study
* Willing to consent to the study
* Male or female who is either post-menopausal, surgically sterile, or if has a childbearing potential, a negative pregnancy test within 2 days prior to the MRI study.

Exclusion Criteria:

* Renal dysfunction (estimated glomerular filtration rate < 60 mL/min/1.73m2) within 6 months
* Metallic implants, pacemaker, blood vessel clip (contra-indicated for MRI)
* Patient size exceeds MRI bore/table limits: (Max body diameter > 60 cm, weight > 136 kg)
* History of gadolinium contrast allergy or intolerance
* Second or third degree AV block
* Sinus node dysfunction
* Acute myocardial infarction (past 3 months)
* Actively wheezing or with acute asthma or bronchospastic attacks requiring changes in therapy within the past 30 days
* Patients that have experienced a previous hypersensitivity reaction thought to be related to regadenoson

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Bateman, MD, Principal Investigator — Aspire Foundation
Locations (1):
- Saint Luke's Health System, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from two groups: a population with coronary artery disease (CAD) of those with low-likelihood-CAD (Control). The myocardial segment perfusion and wall motion scores from the prior clinical positron-emission-tomography (PET) were used to classify segments as one of the following: CONTROL, CAD_REMOTE, CAD_REVERSIBLE.
Pre-assignment Details: Cardiac Magnetic Resonance (CMR) imaging was performed in the same order for all subjects with rest imaging preceding regadenoson stress imaging.
  The same prescription for tagged CMR slice locations (basal, mid, and apical) were used at both rest and stress.
Groups:
- CONTROL: Myocardial strain imaging was performed for all subjects in a similar order. Rest-tag imaging was performed first, then Stress-tag imaging was performed at maximal heart rate following administration of the regadenoson dose.
  Strain values were then calculated for each of 16-segments for each subject. Segments are classified based on myocardial perfusion imaging scores.
  A Control subject is an individual from a population of low-likelihood CAD exhibiting both normal perfusion score and normal wall motion score rest-to-stress as indicated on a clinically indicated PET.
- Coronary Artery Disease: Myocardial strain imaging was performed for all subjects in a similar order. Rest-tag imaging was performed first, then Stress-tag imaging was performed at maximal heart rate following administration of the regadenoson dose.
  Strain values were then calculated for each of 16-segments for each subject. Segments are classified based on myocardial perfusion imaging scores.
  A Coronary Artery Disease (CAD) subject is an individual from a population with CAD exhibiting both normal perfusion and normal wall motion scores (rest-to-stress) on a prior clinically indicated PET.
Period: Overall Study
Arm/Group | CONTROL | Coronary Artery Disease
Started (03SEPT2014) | 15 (Number of subjects recruited for the CONTROL group.) | 25 (Number of subjects recruited for the CAD group.)
Completed (16JAN2018) | 13 (Number of subjects recruited to the Control group meeting all inclusion criteria.) | 23 (Number of subjects recruited to the CAD group meeting all inclusion criteria.)
Not Completed | 2 | 2
Not completed — Safety Screening | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- CONTROL: Myocardial strain imaging was performed for all subjects in a similar order. Rest-tag imaging was performed first, then Stress-tag imaging was performed at maximal heart rate following administration of the regadenoson dose.
  Strain values were then calculated for each of 16-segments for each subject. Segments are classified based on myocardial perfusion imaging scores.
  A control subject is an individual from a low-likelihood CAD population with a prior clinically indicated PET with perfusion and wall motion scores (rest-to-stress).
- Coronary Artery Disease: Myocardial strain imaging was performed for all subjects in a similar order. Rest-tag imaging was performed first, then Stress-tag imaging was performed at maximal heart rate following administration of the regadenoson dose.
  Strain values were then calculated for each of 16-segments for each subject. Segments are classified based on myocardial perfusion imaging scores.
  A Coronary artery disease subject is an individual from a CAD population with a prior clinically indicated PET with perfusion and wall motion scores (rest-to-stress).
- Total: Total of all reporting groups
Arm/Group | CONTROL | Coronary Artery Disease | Total
Number analyzed (Participants) | 13 | 23 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10) | 72 (9) | 66 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 4 | 16 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32 (6) | 31 (6) | 31 (6)

OUTCOME MEASURES:

1. Primary Outcome: RADIAL STRAIN
Description: A measurement of the relative displacement between myocardial points between end-diastole and end-systole along a common ray extending from the center of the left ventricular (LV) cavity (analogous to myocardial thickening). A normal radial strain is indicated by a positive decimal value and can be understood as the percentage change in wall thickness of a myocardial segment. A POSITIVE change in radial strain indicates an increase in wall thickening.
  Because strain is a measurement in change in length (distance) divided by an original length (distance) it is considered unitless.
Time Frame: Day 1
Population: Myocardial segments classified according to subject groups and myocardial perfusion and wall motion scores on prior positron-emission-tomography (PET).
Measure: Mean (Standard Deviation); unit: unitless (strain)
Units Other Than Participants: myocardial segments
Groups:
- CONTROL: A myocardial segment from an individual from a low-likelihood coronary-artery-disease (CAD) population exhibiting both normal perfusion and normal wall motion scores (rest-to-stress) on a prior clinically indicated PET.
- CAD_REMOTE: A myocardial segment from an individual from a population with CAD exhibiting normal perfusion scores and normal wall motion scores (rest-to-stress) on a prior clinically indicated PET.
- CAD_REVERSIBLE: A myocardial segment from an individual from a population with CAD exhibiting a change in perfusion scores and a change in wall motion scores (rest-to-stress) on a prior clinically indicated PET.
Arm/Group | CONTROL | CAD_REMOTE | CAD_REVERSIBLE
Number analyzed (Participants) | 13 | 23 | 23
Number analyzed (myocardial segments) | 203 | 159 | 60
unitless (strain)
  REST | 0.158 (0.100) | 0.149 (0.098) | 0.150 (0.094)
  REGADENOSON STRESS | 0.190 (0.113) | 0.167 (0.104) | 0.141 (0.085)
  REST-to-STRESS CHANGE | 0.033 (0.137) | 0.022 (0.107) | -0.009 (0.099)
Statistical Analysis 1: Comparison: CONTROL; REST-TO-REGADENOSON STRESS; Test type: Superiority; p = 0.001, paired, t-test; non-adjusted
Statistical Analysis 2: Comparison: CAD_REMOTE; REST-TO-REGADENOSON STRESS; Test type: Superiority; p = 0.017, paired, t-test — non-adjusted
Statistical Analysis 3: Comparison: CAD_REVERSIBLE; REST-TO-REGADENOSON STRESS; Test type: Superiority; p = 0.495, paired, t-test — non-adjusted
Statistical Analysis 4: Comparison: CONTROL vs CAD_REMOTE; REST; Test type: Superiority; p = 0.365, t-test, 2 sided; non-adjusted
Statistical Analysis 5: Comparison: CONTROL vs CAD_REVERSIBLE; REST; Test type: Superiority; p = 0.602, t-test, 2 sided; non adjusted
Statistical Analysis 6: Comparison: CAD_REMOTE vs CAD_REVERSIBLE; REST; Test type: Superiority; p = 0.915, t-test, 2 sided; non adjusted
Statistical Analysis 7: Comparison: CONTROL vs CAD_REMOTE; Regadenoson STRESS; Test type: Superiority; p = 0.033, t-test, 2 sided; non adjusted
Statistical Analysis 8: Comparison: CONTROL vs CAD_REVERSIBLE; Regadenoson STRESS; Test type: Superiority; p = 0.002, t-test, 2 sided; non adjusted
Statistical Analysis 9: Comparison: CAD_REMOTE vs CAD_REVERSIBLE; Regadenoson STRESS; Test type: Superiority; p = 0.087, t-test, 2 sided; non adjusted
Statistical Analysis 10: Comparison: CONTROL vs CAD_REMOTE; REST-TO-STRESS CHANGE; Test type: Superiority; p = 0.399, t-test, 2 sided; non adjusted
Statistical Analysis 11: Comparison: CONTROL vs CAD_REVERSIBLE; REST-TO-STRESS Change; Test type: Superiority; p = 0.030, t-test, 2 sided; non adjusted
Statistical Analysis 12: Comparison: CAD_REMOTE vs CAD_REVERSIBLE; REST-TO-STRESS Change; Test type: Superiority; p = 0.048, t-test, 2 sided; non adjusted

2. Primary Outcome: CIRCUMFERENTIAL STRAIN
Description: A measurement of the relative displacement of myocardial points directed along the circumference of the ventricular wall at a given radial distance from the left ventricular (LV) cavity center (e.g. midline). A normal circumferential strain is indicated by a negative decimal value and can be understood as the percentage shortening along the ventricular wall with a greater negative value indicating greater ventricular shortening along the circumference. A positive change in strain would therefore be interpreted as a decrease in circumferential shortening.
  Because strain is a measurement in change in length (distance) divided by an original length (distance) it is considered unitless.
Time Frame: Day 1
Population: Myocardial segments from the population groups according to the AHA 16-segment model and classified according to PET perfusion and wall motion scores.
Measure: Mean (Standard Deviation); unit: strain (unitless)
Units Other Than Participants: myocardial segments
Groups:
- CONTROL: A myocardial segment from an individual from a low-likelihood CAD population exhibiting both normal perfusion and normal wall motion scores (rest-to-stress) on a prior clinically indicated PET.
Arm/Group | CONTROL | CAD_REMOTE | CAD_REVERSIBLE
Number analyzed (Participants) | 13 | 23 | 23
Number analyzed (myocardial segments) | 203 | 159 | 60
strain (unitless)
  REST | -0.181 (0.056) | -0.140 (0.057) | -0.121 (0.054)
  REGADENSOSON STRESS | -0.169 (0.059) | -0.150 (0.053) | -0.126 (0.066)
  REST-to-STRESS CHANGE | 0.012 (0.065) | -0.013 (0.051) | -0.006 (0.051)
Statistical Analysis 1: Comparison: CONTROL; Rest VS Regadenoson Stress; Test type: Superiority; p = 0.011, paired, t-test — Non-adjusted
Statistical Analysis 2: Comparison: CAD_REMOTE; Rest VS Regadenoson Stress; Test type: Superiority; p = 0.003, paired t-test — non-adjusted
Statistical Analysis 3: Comparison: CAD_REVERSIBLE; Rest VS Regadenoson Stress; Test type: Superiority — non-adjusted; p = 0.390, paired, t-test
Statistical Analysis 4: Comparison: CONTROL vs CAD_REMOTE; REST; Test type: Superiority — non-adjusted; p < 0.000, t-test, 2 sided
Statistical Analysis 5: Comparison: CONTROL vs CAD_REVERSIBLE; REST; Test type: Superiority — non-adjusted; p < 0.000, t-test, 2 sided
Statistical Analysis 6: Comparison: CAD_REMOTE vs CAD_REVERSIBLE; REST; Test type: Superiority — non-adjusted; p = 0.022, t-test, 2 sided
Statistical Analysis 7: Comparison: CONTROL vs CAD_REMOTE; Regadenoson STRESS; Test type: Superiority; p = 0.001, t-test, 2 sided — non-adjusted
Statistical Analysis 8: Comparison: CONTROL vs CAD_REVERSIBLE; Regadenoson STRESS; Test type: Superiority; p < 0.000, t-test, 2 sided — non-adjusted
Statistical Analysis 9: Comparison: CAD_REMOTE vs CAD_REVERSIBLE; Regadenoson STRESS; Test type: Superiority; p = 0.006, t-test, 2 sided — non-adjusted
Statistical Analysis 10: Comparison: CONTROL vs CAD_REMOTE; REST-TO-STRESS Change; Test type: Superiority; p < 0.000, t-test, 2 sided; non-adjusted
Statistical Analysis 11: Comparison: CONTROL vs CAD_REVERSIBLE; REST-TO-STRESS Changes; Test type: Superiority; p = 0.058, t-test, 2 sided; non-adjusted
Statistical Analysis 12: Comparison: CAD_REMOTE vs CAD_REVERSIBLE; REST-TO-STRESS Change; Test type: Superiority; p = 0.310, t-test, 2 sided; non-adjusted

3. Secondary Outcome: Late Gadolinium Enhancement (LGE) and RADIAL Myocardial Strain
Description: For each subject, the 16-segments were visually assessed along the short-axis plane for the presence of LGE. These images were collected post regadenoson stress recovery using an inversion-recovery prepared, fast gradient echo sequence and a delay of at least 8 minutes after administration of a single dose of gadobenate dimeglumine.
  The presence of LGE within a segment is a separate classification of segment type. The segment classifications in the other outcomes are determined from the prior positron-emission-tomography (PET) examination where the LGE determination is based solely on cardiac magnetic resonance (CMR) imaging collected data.
  The measurement was performed to determine if the presence of LGE within a particular segment affect the resulting strain?
Time Frame: Day 1
Population: LGE imaging by CMR was acquired only in subjects meeting GFR restrictions.
Measure: Mean (Standard Deviation); unit: strain (unitless)
Units Other Than Participants: Myocardial Segments
Groups:
- LGE-: A myocardial segment from an individual from a population with CAD exhibiting normal perfusion scores and normal wall motion scores (rest-to-stress) on a prior clinically indicated PET.
- LGE+: A myocardial segment from an individual from a population with CAD exhibiting a change in perfusion scores and a change in wall motion scores (rest-to-stress) on a prior clinically indicated PET.
Arm/Group | CONTROL | LGE- | LGE+
Number analyzed (Participants) | 13 | 23 | 23
Number analyzed (Myocardial Segments) | 208 | 143 | 17
strain (unitless)
  REST | 0.157 (0.100) | 0.155 (0.097) | 0.140 (0.074)
  REGADENOSON STRESS | 0.190 (0.113) | 0.185 (0.107) | 0.132 (0.091)
  REST-to_STRESS | 0.032 (0.136) | 0.031 (0.116) | -0.008 (0.089)
Statistical Analysis 1: Comparison: CONTROL; REST vs STRESS; Test type: Superiority; p = 0.001, paired, t-test; non adjusted
Statistical Analysis 2: Comparison: LGE-; REST vs STRESS; Test type: Superiority; p = 0.002, paired, t-test; non adjusted
Statistical Analysis 3: Comparison: LGE+; REST vs STRESS; Test type: Superiority; p = 0.721, paired, t-test; non adjusted
Statistical Analysis 4: Comparison: CONTROL vs LGE-; REST; Test type: Superiority; p = 0.797, t-test, 2 sided; non adjusted
Statistical Analysis 5: Comparison: CONTROL vs LGE+; REST; Test type: Superiority; p = 0.474, t-test, 2 sided; non adjusted
Statistical Analysis 6: Comparison: LGE- vs LGE+; Test type: Superiority; p = 0.537, t-test, 2 sided; non adjusted
Statistical Analysis 7: Comparison: CONTROL vs LGE-; Regadenoson STRESS; Test type: Superiority; p = 0.717, t-test, 2 sided; non adjusted
Statistical Analysis 8: Comparison: CONTROL vs LGE+; Regadenoson STRESS; Test type: Superiority; p = 0.041, t-test, 2 sided; non adjusted
Statistical Analysis 9: Comparison: LGE- vs LGE+; Regadenoson STRESS; Test type: Superiority; p = 0.050, t-test, 2 sided; non adjusted
Statistical Analysis 10: Comparison: CONTROL vs LGE-; REST-to-STRESS Change; Test type: Superiority; p = 0.908, t-test, 2 sided — non adjusted
Statistical Analysis 11: Comparison: CONTROL vs LGE+; Test type: Superiority; p = 0.233, t-test, 2 sided; non adjusted
Statistical Analysis 12: Comparison: LGE- vs LGE+; REST-to-STRESS Change; Test type: Superiority; p = 0.187, t-test, 2 sided; non adjusted

4. Secondary Outcome: Adverse Events
Description: Adverse events were monitored and recorded on a specific Adverse Event (AE) log.
Time Frame: Day 1
Population: Count of Adverse Events not clinically expect and reportable to IRB.
Measure: Count of Participants; unit: Participants
Groups:
- Regadenoson: Regadenoson is a single-use, pre-filled syringe containing 0.4 mg/5 mL of regadenoson.
  Regadenoson: Regadenoson injection is a pharmacologic stress agent indicated for radionuclide myocardial perfusion imaging.
  All subjects received a dose of Regadenoson to perform stress imaging of myocardial strain within a single cardiac magnetic resonance (CMR) imaging session.
Arm/Group | Regadenoson
Number analyzed (Participants) | 36
Participants
  No Adverse Events | 7
  Adverse Events | 29
  Serious Adverse Events | 0

5. Secondary Outcome: Late Gadolinium Enhancement and CIRCUMFERENTIAL Myocardial Strain
Description: The Effects of the presence of LGE on CIRCUMFERENTIAL myocardial Strain
Time Frame: Day 1
Population: LGE as determined by CMR imaging using the AHA 16 segment model.
Measure: Mean (Standard Deviation); unit: strain (unitless)
Units Other Than Participants: Myocardial Segments
Arm/Group | CONTROL | LGE- | LGE+
Number analyzed (Participants) | 13 | 160 | 160
Number analyzed (Myocardial Segments) | 208 | 143 | 17
strain (unitless)
  REST | -0.181 (0.057) | -0.139 (0.052) | -0.101 (0.063)
  REGADENOSON STRESS | -0.169 (0.059) | -0.150 (0.052) | -0.111 (0.051)
  REST-to-STRESS | 0.012 (0.066) | -0.011 (0.046) | -0.010 (0.051)
Statistical Analysis 1: Comparison: CONTROL; REST vs STRESS; Test type: Superiority; p = 0.008, paired, t-test; non adjusted
Statistical Analysis 2: Comparison: LGE-; REST vs STRESS; Test type: Superiority; p = 0.006, paired, t-test; non adjusted
Statistical Analysis 3: Comparison: LGE+; REST vs STRESS; Test type: Superiority; p = 0.428, paired, t-test; non adjusted
Statistical Analysis 4: Comparison: CONTROL vs LGE-; REST; Test type: Superiority; p < 0.000, t-test, 2 sided; non adjusted
Statistical Analysis 5: Comparison: CONTROL vs LGE+; REST; Test type: Superiority; p < 0.000, t-test, 2 sided; non adjusted
Statistical Analysis 6: Comparison: LGE- vs LGE+; REST; Test type: Superiority; p = 0.006, t-test, 2 sided; non adjusted
Statistical Analysis 7: Comparison: CONTROL vs LGE-; Regadenoson STRESS; Test type: Superiority; p = 0.002, t-test, 2 sided; non adjusted
Statistical Analysis 8: Comparison: CONTROL vs LGE+; Regadenoson STRESS; Test type: Superiority; p < 0.000, t-test, 2 sided; non adjusted
Statistical Analysis 9: Comparison: LGE- vs LGE+; Regadenoson STRESS; Test type: Superiority; p = 0.004, t-test, 2 sided; non adjusted
Statistical Analysis 10: Comparison: CONTROL vs LGE-; REST-to-STRESS Change; Test type: Superiority; p < 0.000, t-test, 2 sided; non adjusted
Statistical Analysis 11: Comparison: CONTROL vs LGE+; REST-to-STRESS Change; Test type: Superiority; p = 0.172, t-test, 2 sided; non adjusted
Statistical Analysis 12: Comparison: LGE- vs LGE+; REST-to-STRESS Change; Test type: Superiority; p = 0.957, t-test, 2 sided; non adjusted

ADVERSE EVENTS:
Time Frame: Day 1
Groups:
- Regadenoson: Regadenoson is a single-use, pre-filled syringe containing 0.4 mg/5 mL of regadenoson.
  Regadenoson: Regadenoson injection is a pharmacologic stress agent indicated for radionuclide myocardial perfusion imaging.
  Strain imaging was performed on ALL subjects in the same order with resting strain preceding regadenoson stress strain. Myocardial segments were classified based on prior clinical positron-emission-tomography (PET) results so that segmental strain response to regadenoson could be observed.
Arm/Group | Regadenoson
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 29/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regadenoson (N=36)
Dyspnea (General disorders) | 11
Chest Discomfort (General disorders) | 10
Headache (General disorders) | 8
Flushing (General disorders) | 7
Abdominal: ache/discomfort (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Numbness: Jaw/shoulder (General disorders) | 4
Anxiety (General disorders) | 3
Palpitations (Cardiac disorders) | 2

LIMITATIONS AND CAVEATS:
Reported strain is not adjusted for myocardial mass.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT02115308/Prot_SAP_000.pdf